CLINICAL TRIAL: NCT07318805
Title: A PHASE 1 DOSE ESCALATION AND EXPANSION STUDY TO EVALUATE SAFETY, TOLERABILITY, PHARMACOKINETICS, PHARMACODYNAMICS, AND ANTI-TUMOR ACTIVITY OF PF-08032562 IN PARTICIPANTS WITH ADVANCED OR METASTATIC SOLID TUMORS
Brief Title: A Study to Learn About the Study Medicine Called PF-08032562 in People With Advanced or Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: C6321001
Record Dates: First submitted 2025-12-04; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Advanced Breast Cancer; Metastatic Breast Cancer (HR+/ HER2-); Colorectal Cancer; Metastatic Colorectal Adenocarcinoma; Triple Negative Breast Cancer
Keywords: Carcinoma, Breast; Estrogen Receptor Positive Breast Cancer; HER2- Breast Cancer; Triple Negative Breast Cancer; Colon Cancer
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Triple Negative Breast Neoplasms; Colonic Neoplasms | interventions — Fulvestrant; Cetuximab; Fluorouracil; Oxaliplatin; Leucovorin; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Part 1 Dose Escalation Cohort 1A (Experimental): PF-08032562 monotherapy dose escalation for participants with advanced or metastatic BC or CRC, at different doses and/or schedules of the study drug
  Interventions: Drug: PF-08032562
- Part 1 Dose Escalation Cohort 1B (Experimental): Combination (PF-08032562 + fulvestrant) dose escalation for participants with advanced or metastatic BC, at different doses and/or schedules of the study drug
  Interventions: Drug: PF-08032562; Drug: Fulvestrant
- Part 1 Dose Escalation Cohort 1C (Experimental): Combination (PF-08032562 + cetuximab) dose escalation for participants with advanced or metastatic CRC, at different doses and/or schedules of the study drug
  Interventions: Drug: PF-08032562; Drug: Cetuximab
- Part 1 Dose Escalation Cohort 1D (Experimental): Combination (PF-08032562 + [FOLFOX + bevacizumab]) dose escalation for participants with advanced or metastatic CRC, at different doses and/or schedules of the study drug
  Interventions: Drug: PF-08032562; Drug: Fluorouracil; Drug: Oxaliplatin; Drug: Leucovorin; Drug: Bevacizumab
- Part 2 Dose Expansion Cohort 2A (Experimental): Combination (PF-08032562 + fulvestrant) dose expansion for participants with advanced or metastatic BC, at different doses and/or schedules of the study drug
  Interventions: Drug: PF-08032562; Drug: Fulvestrant
- Part 2 Dose Expansion Cohort 2B (Experimental): PF-08032562 monotherapy or combination (PF-08032562 + cetuximab) dose expansion for participants with advanced or metastatic CRC, at different doses and/or schedules of the study drug
  Interventions: Drug: PF-08032562; Drug: Cetuximab
- Part 2 Dose Expansion Cohort 2C (Experimental): Combination (PF-08032562 + [FOLFOX + bevacizumab]) dose expansion for participants with advanced or metastatic CRC, at different doses and/or schedules of the study drug
  Interventions: Drug: PF-08032562; Drug: Fluorouracil; Drug: Oxaliplatin; Drug: Leucovorin; Drug: Bevacizumab

INTERVENTIONS:
Drug: PF-08032562 — Taken by mouth (PO)
Drug: Fulvestrant — Selective Estrogen Receptor Degrader (SERD)
  Other Names: Faslodex
  Arms: Part 1 Dose Escalation Cohort 1B; Part 2 Dose Expansion Cohort 2A
Drug: Cetuximab — Monoclonal antibody (EGFR inhibitor)
  Other Names: Erbitux
  Arms: Part 1 Dose Escalation Cohort 1C; Part 2 Dose Expansion Cohort 2B
Drug: Fluorouracil — Part of FOLFOX chemotherapy regimen cytotoxic chemotherapy (antimetabolite and pyrimidine analog)
  Other Names: 5-FU; 5-Fluorouracil
  Arms: Part 1 Dose Escalation Cohort 1D; Part 2 Dose Expansion Cohort 2C
Drug: Oxaliplatin — Part of FOLFOX chemotherapy regimen platinum based compound (alkylating agent)
  Other Names: Eloxatin
  Arms: Part 1 Dose Escalation Cohort 1D; Part 2 Dose Expansion Cohort 2C
Drug: Leucovorin — Part of FOLFOX chemotherapy regimen (folic acid analog)
  Other Names: Folinic Acid; Wellcovorin; Calcium Folinate
  Arms: Part 1 Dose Escalation Cohort 1D; Part 2 Dose Expansion Cohort 2C
Drug: Bevacizumab — Monoclonal antibody (VEG-F inhibitor)
  Other Names: Zirabev; Avastin
  Arms: Part 1 Dose Escalation Cohort 1D; Part 2 Dose Expansion Cohort 2C

SUMMARY:
The purpose of this study is to learn about the safety and effects of the study medicine when given alone or together with other anti-cancer therapies. Anti-cancer therapy is a type of treatment to stop the growth of cancer. This study also aims to find the best amount of study medication.

This study is seeking participants that have advanced or metastatic breast cancer (BC), or advanced or metastatic colorectal cancer (CRC).

All participants in this study will take the study medication (PF-08032562) as pill by mouth. This will be repeated for 28-day cycles.

Depending on which part of the study participants are enrolled into, they will receive the study medication PF-08032562 alone or in combination with other anti-cancer medications. The study medication (PF-08032562) will be taken by mouth (PO) in combination with other anti-cancer medications given in the study clinic by intramuscular (IM) injection into the muscle or intravenous (IV) infusion that is directly injected into the veins at different times (depending on the treatment) during the 28-day cycle. The study may also test different schedules.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Advanced or metastatic cancer of the breast or colon Part 1A: metastatic or advanced breast cancer or colorectal cancer for which no standard therapy is available Part 1B: metastatic or advanced breast cancer with disease progression after at least 1 line of treatment with an endocrine therapy and CDK4/6 inhibitor in the advanced or metastatic setting Part 1C: metastatic or advanced colorectal cancer with at least having received chemotherapy and/or targeted therapy if appropriate Part 1D: metastatic or advanced colorectal cancer without any prior chemotherapy for advanced or metastatic disease Part 2A: metastatic or advanced breast cancer with disease progression after at least 1 prior line of CDK4/6 inhibitor and at least 1 prior line of endocrine therapy Part 2B: metastatic or advanced colorectal cancer with at least having received chemotherapy and/or targeted therapy if appropriate Part 2C: metastatic or advanced colorectal cancer without any prior chemotherapy for advanced or metastatic disease
* Measurable disease
* ECOG performance status 0 or 1

Exclusion Criteria:

* Active malignancy within 3 years prior to enrollment
* Known symptomatic brain metastases requiring steroids
* Advanced/metastatic, symptomatic, visceral spread, that are at risk of life-threatening complications in the short term
* Prior irradiation to >25% of the bone marrow
* Hypertension that cannot be controlled by optimal medical therapy
* Renal impairment
* Hepatic dysfunction
* Cardiac abnormalities
* Active bleeding disorder
* Active or history of clinically significant GI disease
* Other unacceptable abnormalities as defined by protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2025-12-16 (Actual); Primary Completion 2029-04-14 (Estimated); Study Completion 2030-04-14 (Estimated)

PRIMARY OUTCOMES:
Part 1 (Dose Escalation): Number of participants with Dose-Limiting Toxicities (DLT) | Baseline up to 28 days
  Any adverse events that are attributable to one, the other, or both study treatments, occurring in the DLT observation period are considered DLTs, excluding toxicities clearly due to underlying disease or extraneous causes.
Part 1 (Dose Escalation): Number of participants with laboratory abnormalities | From start of treatment up to 30 days after last dose or start of new anticancer therapy, whichever occurred first
  Number of participants with laboratory test abnormalities.
Part 1 (Dose Escalation): Incidence of Adverse Events (AEs) | From start of treatment up to 30 days after last dose or start of new anticancer therapy, whichever occurred first
  An adverse event (AE) was any untoward medical occurrence in a participant who received study medication without regard to possibility of causal relationship to it.
Part 2 (Dose Expansion): Objective Response Rate (ORR) | Baseline and every 8 to 12 weeks through time of confirmed disease progression, death, unacceptable toxicity, or through study completion (approximately 2 years)
  ORR defined as per Response Evaluation Criteria in Solid Tumors (RECIST v1.1).

SECONDARY OUTCOMES:
Part 1 & Part 2: Maximum Observed Serum Concentration (Cmax) | Baseline through end of Cycle 1 (each cycle is 28 days)
  Evaluate the single and multiple dose PK of PF-08032562 as monotherapy, or in combination with other anti-tumor agents.
Part 1 & Part 2: Time to Reach Maximum Observed Serum Concentration (Tmax) | Baseline through end of Cycle 1 (each cycle is 28 days)
  Evaluate the single and multiple dose PK of PF-08032562 as monotherapy, or in combination with other anti-tumor agents.
Part 1: Area Under the Curve (AUC) from Time Zero to Last Quantifiable Concentration (AUClast) | Baseline through end of Cycle 1 (each cycle is 28 days)
  Evaluate the single and multiple dose PK of PF-08032562 as monotherapy, or in combination with other anti-tumor agents.
Part 1: Effect of Food on Cmax | Baseline through end of Cycle 1 (each cycle is 28 days)
  Evaluate the effect of food on Cmax of PF-08032562 as monotherapy
Part 1: Effect of Food on Tmax | Baseline through end of Cycle 1 (each cycle is 28 days)
  Evaluate the effect of food on Tmax of PF-08032562 as monotherapy
Part 1: Effect of Food on AUClast | Baseline through end of Cycle 1 (each cycle is 28 days)
  Evaluate the effect of food on AUClast of PF-08032562 as monotherapy
Part 1: Percent change of immune cells within tumors based on immunohistochemistry assessment | Baseline through end of Cycle 1 (each cycle is 28 days)
  Evaluate the single and multiple dose pharmacodynamics of PF-08032562 as monotherapy, or in combination with other anti-tumor agents. This measure will assess change in the concentration of immune cell-related cytokines and chemokines as potential pharmacodynamic effects of PF-08032562 using Immunohistochemistry (IHC) assays.
Part 2 (Dose Expansion): Number of participants with laboratory abnormalities | From start of treatment up to 30 days after last dose or start of new anticancer therapy, whichever occurred first
  Number of participants with laboratory test abnormalities.
Part 2 (Dose Expansion): Incidence of Adverse Events (AEs) | From start of treatment up to 30 days after last dose or start of new anticancer therapy, whichever occurred first
  An adverse event (AE) was any untoward medical occurrence in a participant who received study medication without regard to possibility of causal relationship to it.
Part 1 & Part 2: Objective Response Rate (ORR) as per Response Evaluation Criteria in Solid Tumors (RECIST v1.1) | Baseline and every 8 to 12 weeks through time of confirmed disease progression, death, unacceptable toxicity, or through study completion (approximately 2 years)
  ORR is defined as the percentage of participants in the analysis population having a best overall response (BOR) of confirmed complete response (CR) or confirmed partial response (PR) according to RECIST v1.1.
Part 1 & Part 2: Disease Control Rate (DCR) as per RECIST v1.1 | Baseline and every 8 to 12 weeks through time of confirmed disease progression, death, unacceptable toxicity, or through study completion (approximately 2 years)
  DCR is defined as the proportion of participants with CR or PR with confirmation, or Stable Disease (SD) per RECIST version 1.1.
Part 1 & Part 2: Clinical Benefit Rate (CBR) as per RECIST v1.1 | Baseline and every 8 to 12 weeks through time of confirmed disease progression, death, unacceptable toxicity, or through study completion (approximately 2 years)
  CBR is defined as the percentage of participants with a best overall response of CR or PR at any time before Progressive Disease (PD), or non-CR/non-PD or SD for at least 24 weeks from start date of treatment and prior to PD, relative to the appropriate analysis set.
Part 1 & Part 2: Duration of Response (DOR) as per RECIST v1.1 | Baseline and every 8 to 12 weeks through time of confirmed disease progression, death, unacceptable toxicity, or through study completion (approximately 2 years)
  DOR is defined as the time from first documentation of CR or PR to date of first documentation of PD or death due to any cause.
Part 1 & Part 2: Progression-Free Survival (PFS) as per RECIST v1.1 | Baseline and every 8 to 12 weeks through time of confirmed disease progression, death, unacceptable toxicity, or through study completion (approximately 2 years)
  PFS is defined as time from start date of treatment to the date of first documentation of PD or death due to any cause.
Part 1 & Part 2: Time to Response (TTR) as per RECIST v1.1 | Baseline and every 8 to 12 weeks through time of confirmed disease progression, death, unacceptable toxicity, or through study completion (approximately 2 years)
  TTR is defined as the time from start date of treatment to first documentation of CR or PR.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- United States (3):
  - START Midwest, LLC, Grand Rapids, Michigan
  - START San Antonio, San Antonio, Texas
  - START Mountain Region, West Valley City, Utah

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C6321001